CLINICAL TRIAL: NCT01732172
Title: Study of the Prevalence of a Chronic Inflammatory Condition of the Male Genital Tract at a Distance and Urethritis Following.
Brief Title: Chronic Inflammatory Condition of the Male Genital Tract
Acronym: URIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P 111004
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Urethritis
Keywords: Urethritis; Prevalence of a chronic inflammatory male genital tract
MeSH Terms: conditions — Urethritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient Group (Experimental): Patient with urethritis
  Interventions: Other: Sperm sample
- Control group (Other): Subjects with no urethritis and no history urogenital infection
  Interventions: Other: Sperm sample

INTERVENTIONS:
Other: Sperm sample — Sperm sample

SUMMARY:
Men following after proven and treated urethritis, looking for signs of chronic genital inflammatory syndrome with oxidative stress.

This group of patients will be compared to a control group with no urethritis and no history of urogenital infection. Monocentric, prospective trial.

Duration of study : one year

DETAILED DESCRIPTION:
The presence of leucospermia in an chronic inflammatory genital tract syndrome leads to an oxidative stress and alterations in sperm parameters. Inflammation also affect the glands of the genital tract. This can eventually leads to male infertility, long after the initial infection. But 10% of men who seek treatment for infertility have such a leucospermia, while it is a potentially treatable cause.

Main aim of this study: Search of development of an inflammatory genital tract syndrome in patients with urethritis proven and treated at 6 months after the end of treatment.This group of patients will be compared to a control group with no urethritis and no history of urogenital infection. Monocentric, prospective trial.

Primary endpoint: Seminal elastase value to 6 months after the end of treatment. (500ng/ml or greater)

Secondary objective:

* Search for a genital inflammation in patients with urethritis proven and treated at 12 months after the end of treatment
* Search for oxidative stress in patients with urethritis proven and treated at 6 and 12 months after the end of treatment
* Study of the frequency of relapses infectious and / or passages at the stage of chronic infection after acute urethritis
* Assessment of the parallel evolution of the quality of sperm in the two groups

Progress of research. Time frame Search :

* Duration of inclusions: 12 months
* Duration of patient follow-up: 12 months for control group, 14 months at most for patients taking into account the duration of treatment for urethritis which is 4 to 6 weeks
* Total duration of the study: 26 months

Patients & Methods: French monocentric, prospective trial. 300 subjects are planned to be included for 150 subjects in each group

ELIGIBILITY:
Inclusion criteria common to both groups:

* Subjects aged 18 and over
* Voluntary and signed informed consent

Inclusion criteria specific to the group "patient":

* Patients with clinical signs of urethritis / or
* Patients treated for urethritis following the usual protocols in the month before inclusionand / or
* Patients with positive chlamydial research, or Mycoplasma genitallium or Garderella vaginalis or gonorrhea in the sperm or first urinary stream;

Inclusion criteria specific to the group "control":

- Patients with no urethritis or no history of urogenital infection

Exclusion criteria common to both groups:

* Subjects not wishing to participate in the study
* Subjects that have not signed the informed consent
* Those not affiliated to the social security system (or entitled beneficiary)
* Immunodepressed or have an infection associated with HIV, HBV or HCV
* Chronic systemic disease

Exclusion criteria specific to the group "patient":

- Patients with no signs of urethritis

Exclusion criteria specific to the group "control":

- Subjects with signs of urethritis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2012-12-10 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
Seminal elastase value | 6 months after the end of treatment.
  The dosage of elastase will be do 6 months after the end of treatment.

SECONDARY OUTCOMES:
Seminal elastase value | 12 months after the end of treatment.
  The dosage of elastase will be do 12 months after the end of treatment.
Presence of markers of oxidative stress | 6 to 12 months after the end of treatment
  Presence of markers objectifying the existence of oxidative stress resulting in cellular alterations: Determination of 8-hydroxydeoxyguanosine (8-OHdG) and AOPP (Advanced Oxidation Protein Products)
Functional impairment of the glands of the reproductive tract | 6 to 12 months after the end of treatment
  Presence of biochemical evidence indicating a functional impairment of the glands of the reproductive tract (markers of prostate, seminal vesicles, and epididymis to the seminal biochemistry)
Signs reflecting the sperm function | 6 to 12 months after the end of treatment
  Presence of signs reflecting the sperm function (vitality, mobility, analysis of motion parameters by Computer Assisted Semen Analyzer(CASA))

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe WOLF, MD, PhD, Principal Investigator — Cochin Hospital; Khaled POCATE, MD, Principal Investigator — Cochin Hospital
Locations (1):
- Hospital Cochin, Paris, France